CLINICAL TRIAL: NCT02575963
Title: A Phase I/II Study of Lintuzumab-Ac225 in Older Patients With Untreated Acute Myeloid Leukemia
Brief Title: Lintuzumab-Ac225 in Older Acute Myeloid Leukemia (AML) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: API-01; NCT01756677 (obsolete NCT alias)
Record Dates: First submitted 2015-10-07; First posted 2015-10-15 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: AML
MeSH Terms: interventions — Cytarabine; Furosemide; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phase 1 (Completed) (Experimental): Cytarabine + Lintuzumab-Ac225 Cytarabine days 1 to 10 of each cycle. Doses were divided into 2 equal fractions with the first fraction given approx. 4-7 days after 1 cycle of low dose cytarabine and the second fraction given 4-7 days after the first fraction, followed by up to 11 more cycles. Furosemide (Phase 1 only) and Spironolactone were administered after Lintuzumab-Ac225.
  Experimental: Phase 2
  Experimental: Lintuzumab-Ac225 The Phase II dose determined during the Phase I dose escalation was 4.0 μCi/Kg Lintuzumab-Ac225 and 25 μg/Kg unlabeled HuM195 divided into 2 equal fractions with the first fraction given on Day 1 and the second fraction given on Day 5-8. Spironolactone is administered after Lintuzumab-Ac225.
  Interventions: Drug: Cytarabine (Phase 1 only); Biological: Lintuzumab-Ac225; Drug: Furosemide (Phase 1 only); Drug: Spironolactone

INTERVENTIONS:
Drug: Cytarabine (Phase 1 only) — Low dose cytarabine administered at 20 mg subcutaneously every 12 hours for the first 10 days (Days 1 to 10) of every cycle. Cycle 1 can last up to 52 days (depending on the schedule of study drug dosing) in order to allow for recovery from Lintuzumab-Ac225. Cycles 2-12 will last 28 days each.
  Other Names: Low dose Ara-C; LDAC
Biological: Lintuzumab-Ac225 — In Phase 1 the starting dose level was 1.0 μCi/Kg of Lintuzumab-Ac225 and 15 μg/Kg unlabeled HuM195 divided into 2 equal fractionated doses (0.5 μCi/Kg and 7.5 μg /Kg + 0.5 μCi/Kg and 7.5 μg /Kg) with the first fraction administered approximately 4-7 days after 1 cycle of low dose cytarabine and the second fraction administered 4-7 days after the first fraction, followed by up to 11 more cycles. In Phase 2 the dose will be 4.0 μCi/Kg Lintuzumab-Ac225 and 25 μg/Kg unlabeled HuM195 divided into 2 equal fractions with the first fraction given on Day 1 and the second fraction given on Day 5-8.
  Other Names: HuM195-Ac225; Actimab-A
Drug: Furosemide (Phase 1 only) — 40 mg by mouth daily one day prior to treatment with Lintuzumab-Ac225 and continuing for 10 days following administration of the 2nd divided dose.
  Other Names: Lasix
Drug: Spironolactone — 25 mg by mouth daily, administered 10 days after second dose of 225Ac-HuM195 and continued for 12 months.
  Other Names: Aldactone

SUMMARY:
The study is a multicenter, open label Phase I/II trial.

1. Establish the MTD of fractionated doses of Lintuzumab-Ac225 in combination with low dose cytosine arabinoside (Low Dose Ara-C, LDAC) (Phase 1 portion)
2. Determine the response rate (CR + CRp + CRi) to fractionated doses of Lintuzumab-Ac225 alone (Phase 2 portion)

DETAILED DESCRIPTION:
The study is a multicenter, open label Phase I/II trial. Phase I, dose-escalation: This portion of the overall study uses a 3+3 design to estimate the maximum tolerated dose (MTD). The starting dose level will be 1.0 μCi/Kg of Lintuzumab-Ac225 and 15 μg/Kg unlabeled HuM195 divided into 2 equal fractionated doses (0.5 μCi/Kg and 7.5 μg /Kg + 0.5 μCi/Kg and 7.5 μg /Kg) with the first fraction administered approximately 4 - 7 days after 1 cycle of LDAC (20 mg subQ every 12 h x 10 days administered for cytoreduction) and the second fraction administered 4-7 days after the first fraction. Subjects will then go on to receive up to 11 additional cycles of LDAC or until progression of disease. Three to six patients will be treated at each dose level, and dose escalation will proceed if less than 33% of patients in a cohort experience dose-limiting toxicity.

Phase II, efficacy component. The study was designed as a 2- stage minimax design. Patients will be given two infusions of Lintuzumab-Ac225, 4-8 days apart (Day 5-Day 9), initially at the dose level determined to be the MTD in the Phase I portion. The second dose of Lintuzumab-Ac225 may be delayed up to 14 days after the first dose for clinical or scheduling reasons. Response will be initially assessed on or around days 28-42 after the final study drug administration. The primary endpoint (CR+CRp + CRi) will be determined on day 42. Best response will be evaluated from Day 1, Dose 1 until the end of the study.

ELIGIBILITY:
Phase 1 Major Inclusion Criteria:

1. Untreated AML, including patients with an antecedent hematologic disorder or secondary disease. Patients with prior MDS may have received therapy with immunomodulatory agents or hypomethylating agents for this diagnosis. Patients with other prior cancer diagnoses are allowed as long as they have no measurable disease, are not undergoing active therapy, and have a life expectancy of ≥ 4 months.
2. Patients age ≥60 years who:

   1. Are unwilling to receive intensive (e.g. 7+3) chemotherapy, or
   2. Have poor-risk prognostic factors defined as antecedent hematologic disorder, prior chemotherapy or XRT, abnormal karyotype other than t(8;21), inv16, or t(16;16), any karyotype with FLT3-ITD, or presenting WBC>100K, or
   3. Have significant comorbidities, that in the judgment of the investigator makes the subject unsuitable for standard dose induction chemotherapy (e.g. anthracycline and infusional cytarabine given as 7+3), or;
   4. Any patient age ≥ 70 years.
3. Blast count ≥20%
4. Greater than 25% of blasts must be CD33 positive.
5. Adequate renal and hepatic function
6. ECOG ≤ 3

Phase 2 Inclusion Criteria:

1. Untreated AML, including patients with an antecedent hematologic disorder or secondary disease. Patients with prior MDS may have received therapy with immunomodulatory agents for this diagnosis.
2. Patients age ≥60 years who:

   1. Patients ≥60 years unfit to receive intensive (e.g., 7+3) chemotherapy who have:

      * Congestive heart failure or documented cardiomyopathy with an EF ≤50%, provided that EF ≥35% or,
      * Documented pulmonary disease with DLCO ≤65% or FEV1 ≤65%, provided that patients do not require more than 2 L of oxygen per minute or,
      * Documented liver disease with marked elevation of transaminases >3 x ULN or,
      * Serum creatinine >1.2 mg/dL
   2. Have significant comorbidities, that in the judgment of the investigator makes the subject unsuitable for standard dose induction chemotherapy (e.g., anthracycline and infusional cytarabine given as 7+3); or
   3. Any patient age ≥ 75 years.
3. Blast count ≥ 20% (WHO criteria)
4. Greater than 25% of blasts must be CD33 positive.
5. Have a circulating blast count of less than 200/mm3 (control with hydroxyurea or similar agent is allowed);
6. Creatinine < 2.0 mg/dl
7. Estimated creatinine clearance ≥ 50ml/min
8. Bilirubin ≤ 2.0 mg/dl; AST and ALT < 5.0 times the ULN
9. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2

Exclusion Criteria:

1. Patients with acute promyelocytic leukemia
2. Treatment with chemotherapy or biologic therapy within 3 weeks, except for hydroxyurea, which must be discontinued prior to treatment on study
3. Treatment with radiation within 6 weeks
4. Active serious infections uncontrolled by antibiotics
5. Active malignancy within 2 years of entry, except previously treated non-melanoma skin cancer, carcinoma in situ or cervical intraepithelial neoplasia, and organ confined prostate cancer with no evidence of progressive disease based on PSA levels and are not on active therapy.
6. Clinically significant cardiac or pulmonary disease
7. Patients with liver cirrhosis
8. Active CNS leukemia. Patients with symptoms of CNS involvement, particularly those with M4 or M5 subtypes, should undergo lumbar puncture prior to treatment on study to exclude CNS disease. Symptoms include cranial neuropathies, other neurologic deficits, and headache.
9. Psychiatric disorder that would preclude study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2018-11 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) of Lintuzumab-Ac225 | Cycle 1, up to 52 days
  If two or more patients in a cohort experience dose limiting toxicity (DLT), then maximum tolerated dose (MTD) will have been exceeded, and no further dose escalation will occur. If only three patients were treated at a dose level under consideration as the MTD, then up to three additional patients will be accrued. If no more than one of the six patients at that dose level experiences DLT, then that dose level will be confirmed as the MTD.
Phase II: CR+CRp+CRi | First evaluation at 42 days after treatment
  The primary objective is to determine the antileukemic effects, including its ability to produce complete remissions, of Lintuzumab-Ac225.

SECONDARY OUTCOMES:
Phase II: PFS | 1 year
  Progression Free Survival
Phase II: LFS | 1 year
  Leukemia Free Survival
Phase II: OS | 1 year
  Overall Survival
Phase II: Toxicity Spectrum | 1 year
  Safety Data

CONTACTS AND LOCATIONS:
Overall Officials: Avinash Desai, MD, Study Chair — Actinium Pharmaceuticals Inc.
Locations (17):
- United States (16):
  - UCLA Medical Center, Division of Hematology/Oncology, Los Angeles, California
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - Ochsner Medical Center, The Gayle and Tom Benson Cancer Center, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University Medical, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - St. Francis Cancer Center, Greenville, South Carolina
  - Baylor Scott and White Research Institute, Charles A. Sammons Cancer Center, Dallas, Texas
  - Swedish Cancer Institute, Center for Blood Disorders and Stem Cell Transplantation, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University, Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- VA Caribbean Healthcare System, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larson SM, Carrasquillo JA, Cheung NK, Press OW. Radioimmunotherapy of human tumours. Nat Rev Cancer. 2015 Jun;15(6):347-60. doi: 10.1038/nrc3925. PMID 25998714
- [Background] Jurcic JG, Rosenblat TL. Targeted alpha-particle immunotherapy for acute myeloid leukemia. Am Soc Clin Oncol Educ Book. 2014:e126-31. doi: 10.14694/EdBook_AM.2014.34.e126. PMID 24857092
- [Background] Scheinberg DA, McDevitt MR. Actinium-225 in targeted alpha-particle therapeutic applications. Curr Radiopharm. 2011 Oct;4(4):306-20. doi: 10.2174/1874471011104040306. PMID 22202153
- [Derived] Nikitaki Z, Velalopoulou A, Zanni V, Tremi I, Havaki S, Kokkoris M, Gorgoulis VG, Koumenis C, Georgakilas AG. Key biological mechanisms involved in high-LET radiation therapies with a focus on DNA damage and repair. Expert Rev Mol Med. 2022 Mar 31;24:e15. doi: 10.1017/erm.2022.6. PMID 35357290
- See also: Phase I trial of alpha-particle immunotherapy with 225Ac-lintuzumab and low-dose cytarabine in patients age 60 or older with untreated acute myeloid leukemia. — http://jnm.snmjournals.org/content/58/supplement_1/456.abstract?sid=5073e99e-45a1-42c7-8f12-4d438e4a98d9&utm_source=TrendMD&utm_medium=cpc&utm_campaign=J_Nucl_Med_TrendMD_1
- See also: Phase I Trial of Targeted Alpha-Particle Immunotherapy with Actinium-225 (225Ac)-Lintuzumab (Anti-CD33) and Low-Dose Cytarabine (LDAC) in Older Patients with Untreated Acute Myeloid Leukemia (AML) — https://ash.confex.com/ash/2015/webprogramscheduler/Paper81957.html